CLINICAL TRIAL: NCT04316767
Title: Smartphone Delivery of Cognitive Behavioral Therapy for Post-intensive Care Syndrome-Family: A Pilot Study
Brief Title: Self-care App for Family Members of ICU Patients.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kent State University (Other)
Collaborators: Summa Health System (Other)
Responsible Party: Principal Investigator, Amy Petrinec, Assistant Professor, Kent State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AACN 416051
Record Dates: First submitted 2020-03-17; First posted 2020-03-20 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Post Intensive Care Unit Syndrome
Keywords: PICS-F; mobile health app; health-related quality of life; mental health self-efficacy; cognitive behavioral therapy; ICU family

STUDY DESIGN:
Intervention Model Description: A prospective, repeated measures, longitudinal design with randomization to one of two parallel groups (control, intervention) will be employed. Participants will be randomized to group assignment after study enrollment is completed and baseline measurements are obtained.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- App Intervention (Experimental): Participants will download a mobile self-care app on their smartphones. The app guides users through exercises based on cognitive behavioral therapy principles. Participants will be able to use the app as frequently as desired throughout the course of the study.
  Interventions: Behavioral: App Intervention
- Control (No Intervention): Participants will receive usual supportive care provided to family members of ICU patients.

INTERVENTIONS:
Behavioral: App Intervention — Participants will receive access to a self-care app for use on their smartphone. The app provides a suite of tools based on cognitive behavioral therapy and mindfulness. The app guides users through a variety of short lessons (3-5 minutes) that teach users to self-manage stress, mood, anxiety, and depression. Participants will be encouraged to use the app on a daily basis and will be able to use the app at their discretion.
  Other Names: Sanvello app
  Arms: App Intervention

SUMMARY:
Family members of critically ill (ICU) patients are at risk for developing significant symptoms of anxiety, depression, and post-traumatic stress during and after the ICU experience. Cognitive behavioral therapy is a form of therapy that can help individuals cope with stressful events in a more active and effective way. This study will examine the effectiveness of a smartphone self-care app delivering cognitive behavioral therapy in decreasing the psychological symptoms suffered by ICU family members. Half of the sample will receive the self-care app and half of the study sample will receive the usual supportive care given to family members of ICU patients. The researchers anticipate the self-care app will diminish the severity of anxiety, depression, and post-traumatic stress symptoms experienced by ICU family members.

DETAILED DESCRIPTION:
Family members of critically ill patients suffer symptoms of post-intensive care syndrome-family (PICS-F), including anxiety, depression, and post-traumatic stress disorder with a diminished quality of life. These symptoms persist long after the episode of critical illness and can linger for years. Cognitive behavioral therapy has become the primary non-pharmacological treatment of an increasing list of psychological symptoms and disorders, including anxiety, depression, and post-traumatic stress. For mild-to-moderate symptoms, mobile technology delivery of cognitive behavioral therapy without input from a clinician has been found to be feasible and well-accepted with efficacy that rivals face-to-face therapy.

The purpose of this pilot study is to examine the efficacy of smartphone delivery of cognitive behavioral therapy via a mobile health app (intervention) on the severity and prevalence of PICS-F symptoms in family members of critically ill patients. The study will include family members of critically ill patients admitted to two 26-bed ICUs at the Akron campus of Summa Health System. A prospective, repeated measures, longitudinal design with randomization to two groups (control, intervention) will be employed. Primary outcome measures will include symptoms of PICS-F (anxiety, depression, post-traumatic stress), health-related quality of life, and mental health self-efficacy measured at enrollment, 30 days after enrollment, and 60 days after enrollment. App usage over the course of the study (number of logins, total time spent with app) will be obtained at the final time point of the study (60 days after enrollment). A sample size of 60 family members is planned for this pilot study (30 intervention, 30 control). The sample size was determined according to the recommendations of Whitehead et al.estimating an a priori small effect size and an attrition rate of 30% derived from previous studies.

The aims of the study are:

Aim 1: Determine the prevalence and severity of PICS-F symptoms (anxiety, depression, post-traumatic stress), health-related quality of life (HRQOL), and mental health self-efficacy (MHSE) in family decision makers of critically ill patients and their change over time (enrollment, 30 days, 60 days).

Aim 2: Determine differences in PICS-F symptom severity, HRQOL, and MHSE in family decision makers of critically ill patients receiving a mobile health app (MHapp) intervention compared to family members receiving standard care and support.

Aim 3: Determine the relationship between the dose of the MHapp (total time spent with the app, total log-ins) over the course of the study (60 days) and changes in PICS-F symptom severity (anxiety, depression, post-traumatic stress), HRQOL, and MHSE.

Data Analysis and Statistical Plan: Data will be analyzed using Statistics Package for the Social Sciences (SPSS, Version 25) software. Descriptive statistics will be used to assess frequencies and variability of the data, coding inaccuracies, outliers, and missing data. The statistical plan for each specific aim is as follows:

Aim 1: The investigators will report study variables with descriptive statistics. Change over time will be examined with repeated measures ANOVA.

Aim 2: Differences between intervention and control groups will be assessed with student's t-test. Differences between groups in regard to severity of PICS-F symptoms will be used to calculate effect size for the intervention.

Aim 3: Relationship between total MHapp dose and longitudinal change in study variables will be examined with Pearson's correlation.

Human Subjects and Ethical Issues: The research presents no more than minimal psychological risk or harm, largely from the possibility that answering the questions on the anxiety, depression, and stress instruments may be distressing for participants. Psychological risk will be minimized by emphasizing that study participants can stop participating in the study at any time and are not obligated to answer any question that they find distressing. Family members who endorse clinically significant symptoms will be referred to their primary care physician. Family members of patients who die during the study will be referred to local bereavement support groups.

There is a low risk of privacy or confidentiality loss. Risk will be minimized by the following measures: (a) the only record linking the participant and the research data is the consent document; (b) consent documents will be kept in a locked cabinet in the locked office of the PI; (c) data will be entered and stored by the RA on REDCap, a secure, HIPAA-compliant web-based platform; (d) all data files obtained for analysis will be stored on a password-protected laptop computer stored in a locked room; and (e) The PI, co-investigators, and research assistant (RA) are the only individuals with access to the data files.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* self-identifies as the family decision-maker of the critically ill patient
* reads and speaks English
* owns a smartphone with iOS or Android operating system
* critically ill family member has been in the ICU greater than three days
* critically ill family member is mechanically ventilated and lacks cognitive capacity
* critically ill family member is not expected to be transferred out of the ICU within the next 48 hours
* critically ill family member is 18 years of age or older.

Exclusion Criteria:

* Employee of Summa Health System

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-08-28 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Change in anxiety-Hospital Anxiety and Depression Scale (HADS) | Baseline, 30 days, 60 days
  The HADS is a 14-item self-report scale with seven items forming an anxiety subscale (HADS-A) and seven items forming a depression subscale (HADS-D). Each of the two subscales can have scores ranging from 0-21 with higher scores indicating higher levels of anxiety or depression symptoms.
Change in depression-Hospital Anxiety and Depression Scale (HADS) | Baseline, 30 days, 60 days
  The HADS is a 14-item scale with seven items forming an anxiety subscale (HADS-A) and seven items forming a depression subscale (HADS-D). Each of the two subscales can have scores ranging from 0-21 with higher scores indicating higher levels of anxiety or depression symptoms.
Change in post-traumatic stress measured by the PTSD Checklist for DSM-5 (PCL-5) | Baseline, 30 days, 60 days
  The PCL-5 is a 20-item self-report measure corresponding to the Diagnostic and Statistical Manual of Mental Disorders 5th edition (DSM-5) criteria for PTSD. A total symptom severity score (0-80) can be obtained by summing all of the items with higher scores indicating higher severity of PTSD symptoms.
Change in health-related quality of life measured by Medical Outcomes Study 12-item Short-Form General Health Survey (SF- 12) | Baseline, 60 days
  The SF-12 is a 12-item self-report scale measuring health-related quality of life. Each item on the scale is scored using a Likert-type scale with raw scores transformed to a 0 (worst) to 100 (best) scale. The scale provides a summary score of 0 to 100 for physical and mental quality of life with higher scores representing a more positive quality of life.
Change in Mental Health Self-Efficacy Scale (MHSES) score | Baseline, 30 days, 60 days
  The MHSES is a 6-item scale measuring mental health self-efficacy. Each item is measured on a 10-point Likert scale ranging from 1 (not at all confident) to 10 (totally confident). Items are summed for a total score ranging from 6-60 with higher scores indicating higher levels of mental health self-efficacy.

SECONDARY OUTCOMES:
App usage | From enrollment to study completion (60 days)
  Total number of logins and total number of minutes spent using app

CONTACTS AND LOCATIONS:
Overall Officials: Amy B Petrinec, PhD, Principal Investigator — Kent State University
Locations (1):
- Summa Health System, Akron, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available.

REFERENCES:
- [Derived] Petrinec AB, Hughes JW, Zullo MD, Wilk C, George RL. Smartphone Delivery of Cognitive Behavioral Therapy for Postintensive Care Syndrome-Family: Protocol for a Pilot Study. JMIR Res Protoc. 2021 Aug 4;10(8):e30813. doi: 10.2196/30813. PMID 34346900